CLINICAL TRIAL: NCT06698146
Title: Colorectal Metastasis to Liver Extraction With Auxiliary Transplant and Delayed Resection Registry Study
Brief Title: Colorectal Metastasis to Liver Extraction With Auxiliary Transplant and Delayed Resection
Acronym: CLEAR
Status: Recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Zachary Dietch, Assistant Professor, Surgery (Organ Transplant), Northwestern University
Other Study IDs: STU00222933
Record Dates: First submitted 2024-11-14; First posted 2024-11-20 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-04

CONDITIONS: Liver Transplant Surgery; Colorectal Cancer Metastatic; Colon Cancer Liver Metastases
Keywords: Liver Transplant; Colorectal Cancer Metastatic; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Living Donor Liver Transplant: Living Donor Liver Transplant using right or left lobe donor graft
- RAPID Living Donor Liver Transplant (using LLS or left lobe): Resection And Partial Liver Transplantation with Delayed Total Hepatectomy is a two staged procedure that utilized partial donor grafts and stages hepatectomies. In the first stage, a left hepatectomy is performed and a LT is performed using a donor left lateral segment split (LLS) (or left lobe split in some circumstances). Once the LT has achieved sufficient volume (typically within two weeks), a right hepatectomy is performed to remove all native liver, leaving the LT intact.
- RAPID Deceased Donor Liver Transplant (LLS or left lobe): Resection And Partial Liver Transplantation with Delayed Total Hepatectomy is a two staged procedure that utilized partial donor grafts and stages hepatectomies. In the first stage, a left hepatectomy is performed and a LT is performed using a donor left lateral segment split (LLS) (or left lobe split in some circumstances). Once the LT has achieved sufficient volume (typically within two weeks), a right hepatectomy is performed to remove all native liver, leaving the LT intact.
- Liver Transplant Deceased Donor (Whole Liver): The whole of the deceased donor liver is used. Livers from deceased donors are allocated to potential recipients according to the MELD (Model for End-Stage Liver Disease) scoring system.

SUMMARY:
Liver transplantation (LT) has become an accepted treatment for selected patients with unresectable liver metastases due to colorectal cancer (CRLM). The goal of this study is to look at and compare the clinical results of all the different approved methods (living vs. Deceased, whole organ vs. Split, one staged vs. Two staged) used to perform a standard liver transplant procedure for recipients with CRLM. Investigators will look at things like different procedure results, recovery in the hospital, and survival rates one year after the transplant. Investigators will also take blood samples from participants to be used in future research. All the transplant methods the investigators are comparing are standard practices approved by the United Network of Organ Sharing (UNOS).

ELIGIBILITY:
Inclusion:

1. All Patients of either gender ≥ 18 years of age who are listed for Liver transplant candidates at Northwestern with liver metastases due to colorectal cancer (CRLM).
2. Subjects must be able to provide informed consent themselves and without the use of a legally authorized representative (LAR), to be determined by the PI or Sub-I at the time of Consent.

Exclusion:

1. Adults unable to consent
2. Pregnant Women
3. Certain clinical/surgical/anatomical parameters, at the discretion of the PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Northwestern University participants with liver metastases due to colorectal cancer (CRLM) who are eligible to liver transplant candidates
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2034-01-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Graft and Patient Survival Outcomes | From liver transplant to 12 months
  Graft survival will be measured as the time from transplantation to graft failure, or re-transplantation date.

SECONDARY OUTCOMES:
Outcomes of liver transplant recipients | From liver transplant to 12 months
  Evaluate outcomes (e.g., complications or surgical outcomes) of liver transplant (LT) recipients.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University-Comprehensive Transplant Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No